CLINICAL TRIAL: NCT03647865
Title: Evaluation of The Accuracy of CAD-CAM Custom Made Titanium Miniplates In Positioning of the Genial Segment in Computer Guided Genioplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Nazih Zaki Sedrak, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018
Record Dates: First submitted 2018-05-19; First posted 2018-08-27 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Macrogenia; Microgenia; Miniplate
Keywords: Computer Guided,; Osseous Genioplasty; Custom Made Titanium Plates; Orthognathic Surgery; Genioplasty; patient Specific device

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients need genioplasty (Experimental)
  Interventions: Procedure: Osseous Genioplasty

INTERVENTIONS:
Procedure: Osseous Genioplasty — Surgical Procedure that cuts the chin and reposition it in the correct place

SUMMARY:
In patients with chin deformeties, will using a custom made titanium plate in the positioning of the genial segments give an accurate results in comparison to the preoperative planned osteotomy and move of the Genioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients with genial deformeties that require surgical correction.
* Patients with chin asymmetry.
* Patients older than 18 years old.

Exclusion Criteria:

* Patients with uncontrolled systemic disease (Diabetes Mellitus).
* Previous Radiotherapy to the area of interest.
* Patients on bisphosphonates therapy.
* Patients underwent previous or concomitant mandibular orthognathic surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy Of the Custom Made Miniplate | one year
  Hausdorff function analysis (Topographic Color Mapping) by superimposition of both preoperative and postoperative computed tomography 3D scans and obtaining numerical values.
  Data management and analysis will be performed using Statistical Package for Social Sciences (SPSS) vs.21. Numerical data will be summarized using means and standard deviations or median and range as appropriate. Correlation analysis between Accuracy of computer assisted custom made plate and preoperative 3D virtual planning will be done using Pearson or Sperman rho as appropriate. Paired t test will be done and equivelance limit will be tested. All p- values are two sided. P- Values <0.05 will be considered significant.

SECONDARY OUTCOMES:
Patient Satisfaction (Esthetics) | one year
  Questionnaire with numerical scale ranging from minimal score ( number 1) to maximum score (number 10) in ascending manner where the minimal score indicated unpleasant or unsatisfactory result ( doesn't meet the patient expectation) and maximum score indicated satisfactory and pleasant result (fully meets patient satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Nader Na Elbokle, Phd Holder, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No